CLINICAL TRIAL: NCT02539290
Title: Preovulatory Uterine Flushing With Saline as a Treatment for Unexplained Infertility: A Randomised Controlled Trial Protocol
Brief Title: Preovulatory Uterine Flushing With Saline as a Treatment for Unexplained Infertility
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Quebec-Universite Laval (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2015-1146
Record Dates: First submitted 2015-08-26; First posted 2015-09-03 (Estimated); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Unexplained Infertility; Infertility
Keywords: Unexplained infertility; Infertility; Tubal flushing; Uterine flushing; Live birth; Pregnancy; Randomized controlled trial; Saline; Physiological saline
MeSH Terms: conditions — Infertility | interventions — Sex

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Uterine flushing (Experimental): Detection of ovulation, injection of 20 millilitres of physiological saline by an intra-uterine catheter the day of the luteinizing hormone surge, and sexual intercourse within 12 hours after intervention
  Interventions: Behavioral: Detection of ovulation; Procedure: Uterine flushing; Behavioral: Sexual intercourse
- Vaginal flushing (Sham Comparator): Detection of ovulation, injection of 10 millilitres of physiological saline intravaginally the day of the luteinizing hormone surge, and sexual intercourse within 12 hours after intervention
  Interventions: Behavioral: Detection of ovulation; Procedure: Vaginal flushing; Behavioral: Sexual intercourse

INTERVENTIONS:
Behavioral: Detection of ovulation — Detecting the luteinizing hormone surge using test sticks in a urine sample
Procedure: Uterine flushing — Injection of 20 millilitres of physiological saline by an intra-uterine catheter the day of the luteinizing hormone surge
  Other Names: Tubal flushing
  Arms: Uterine flushing
Procedure: Vaginal flushing — Injection of 10 millilitres of physiological saline intravaginally the day of the luteinizing hormone surge
  Arms: Vaginal flushing
Behavioral: Sexual intercourse — Sexual intercourse on the day of the intervention and the following day

SUMMARY:
The purpose of this study is to determine whether preovulatory uterine flushing with physiological saline is effective in the treatment of unexplained infertility.

DETAILED DESCRIPTION:
In vitro fertilisation is the only current reasonable treatment for unexplained infertility. Uterine flushing, associated with a five-fold increase in pregnancy when performed preovulatory, has been proposed as a new alternative. This treatment could flush out debris or alter inflammatory factors preventing fertilisation and implantation. The objective of this study is to assess the efficacy of pre-ovulatory uterine flushing with physiological saline for the treatment of unexplained infertility. This study is a randomised controlled trial based on consecutive women aged between 18 and 37 years consulting for unexplained infertility for at least one year. The day of their luteinizing hormone surge, 192 participants will be randomised in two equal groups to either receive 20 millilitres of physiological saline by an intra-uterine catheter or 10 millilitres of saline intravaginally. Investigators will assess relative risk of live birth (primary outcome), as well as pregnancy over one cycle of treatment. Side effects, complications, and acceptability of the intervention will be reported.

ELIGIBILITY:
Inclusion Criteria:

* Primary or secondary infertility ≥12 months.
* Diagnosis of unexplained infertility ≤24 months:

  * Anti-Mullerian hormone ≥0.4 ng/mL and/or follicle-stimulating hormone ≤13 IU/L in early follicular phase;
  * regular cycle of 21-35 days,
  * positive ovulation tests, and/or
  * luteal phase serum progesterone ≥25mmol/L in a natural cycle;
  * semen analysis with total motile sperm count ≥ 5 million;
  * normal uterine cavity;
  * patent tubes.
* Negative genitourinary test for gonorrhoea and chlamydia ≤12 months.

Exclusion Criteria:

* Body mass index ≥35 kg/m2.
* Ongoing pregnancy.

Ages: 18 Years to 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 192 (Estimated)
Dates: Start 2015-12-30 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with a live birth resulting from one cycle of treatment | 10 months after randomisation
  Proportion of participants with a live birth resulting from one cycle of treatment based on questionnaire and medical data.

SECONDARY OUTCOMES:
Proportion of participants with a pregnancy resulting from one cycle of treatment | One month after randomisation
  Proportion of participants with a positive urinary or serum pregnancy test, gestational sac on ultrasound or histological evidence of trophoblastic tissue resulting from one cycle of treatment based on questionnaire and medical data.
Adverse effects | One month after randomisation
  Number of participants with treatment-related pain, vagal symptoms, nausea, vomiting, temperature, pelvic infection
Proportion of participants who find the intervention acceptable | One month after randomisation
  Proportion of participants that would be willing to receive the intervention for a second time and find the intervention acceptable.

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie Dodin, MD-MSc, Study Director — Centre Hospitalier Universitaire de Quebec
Locations (1):
- Centre Hospitalier Universitaire de Quebec, Québec, Canada

REFERENCES:
- [Derived] Maheux-Lacroix S, Dodin S, Moore L, Bujold E, Lefebvre J, Bergeron ME. Preovulatory uterine flushing with saline as a treatment for unexplained infertility: a randomised controlled trial protocol. BMJ Open. 2016 Jan 6;6(1):e009897. doi: 10.1136/bmjopen-2015-009897. PMID 26739737